CLINICAL TRIAL: NCT07314073
Title: A Phase 2, Open-label, Non-randomized, Single Center Study Evaluating 18F-Fluoroestradiol Positron Emission Tomography/Computed Tomography for the Detection of Distant Metastases in Low-grade, Estrogen Receptor-positive Stage III Breast Cancer
Brief Title: [18F]FES PET/CT for the Detection of Distant Metastasis in Low-grade ER-positive Stage III Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyehyun Jeong, Assistant professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FES LABC
Record Dates: First submitted 2025-12-03; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Stage III Breast Cancer
Keywords: breast cancer; estrogen receptor; [18F]FES PET/CT; distant metastasis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A phase 2, open-label, non-randomized, single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FES PET/CT (Experimental)
  Interventions: Diagnostic Test: Fluoroestradiol (18F)

INTERVENTIONS:
Diagnostic Test: Fluoroestradiol (18F) — Images for 90 minutes after F-18 FES injection

SUMMARY:
This study aims to evaluate the detection rate of distant metastases using [18F]FES PET/CT in patients with low-grade, ER-positive stage III breast cancer.

DETAILED DESCRIPTION:
Breast cancer is highly prevalent, and approximately 75% of cases are estrogen receptor (ER)-positive. Stage III breast cancer carries a significant risk of distant metastasis; therefore, NCCN and ESMO guidelines recommend systemic staging with CT, bone scan, or 18F-FDG PET/CT. However, 18F-FDG PET/CT demonstrates limited sensitivity in low-grade ER-positive tumors and invasive lobular carcinoma (ILC), and can yield false positives due to inflammatory reaction or reactive hyperplasia. Thus, more accurate imaging modalities are needed in this subgroup.

18F-fluoroestradiol (18F-FES) PET/CT visualizes ER expression and has shown high concordance with histopathology. A phase III study demonstrated 77% sensitivity and 100% specificity for metastatic disease. Emerging evidence suggests that 18F-FES PET/CT may detect distant or regional lymph node metastases more accurately than standard imaging, particularly in ILC and low-grade tumors, and can influence management decisions such as surgery and radiotherapy planning.

Accurate identification of regional nodal involvement (axillary, supraclavicular, internal mammary nodes) is essential for determining the extent of axillary surgery after neoadjuvant chemotherapy and for tailoring regional nodal irradiation. Prior studies show that metabolic imaging can alter radiotherapy fields in up to 40% of patients.

The primary objective is to determine the patient-based detection rate of qualitative 18F-FES PET/CT for distant metastases. Secondary objectives include evaluating its patient-based sensitivity and specificity for distant metastases; determining the detection rate, sensitivity, and specificity for cN3 lymph node metastases (infraclavicular, supraclavicular, and internal mammary nodes); assessing the rate of management change attributable to 18F-FES PET/CT; and comparing 18F-FES PET/CT with 18F-FDG PET/CT for detection rate, diagnostic accuracy, and management impact. Exploratory analyses will examine the correlation between qualitative and quantitative 18F-FES PET/CT findings and pathological response to neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥19 years, regardless of race/ethnicity
2. Patients newly diagnosed with invasive breast cancer within 90 days prior to screening, with documented histopathological confirmation.
3. Patients diagnosed with histologically confirmed estrogen receptor-positive, histologic grade 1 or 2 primary breast cancer
4. Patients with clinical stage IIIA-IIIC disease according to the 8th edition of the American Joint Committee on Cancer (AJCC) TNM staging system
5. Patients who have undergone, or are scheduled to undergo chest computed tomography (CT), abdominal CT, and bone scintigraphy within 90 days prior to screening before the 18F-FES PET/CT scan
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of ≤2

Exclusion Criteria:

* The subject or the subject's legally authorized representative has not signed the informed consent form
* Subjects who are currently receiving systemic therapy for breast cancer (e.g., neoadjuvant chemotherapy, hormonal therapy)
* Subjects with a history of another invasive malignancy within the past 2 years (except for non-melanoma skin cancer)
* Subjects diagnosed with distant metastases on chest CT, abdominal CT, or bone scintigraphy performed within 90 days prior to screening or before the 18F-FES PET/CT scan
* Subjects for whom neither biopsy nor ≥6 months of follow-up imaging has been performed for lesions suspicious for distant metastases
* Pregnant or breastfeeding women. The following cases are considered not at risk of pregnancy: (1) physiologically postmenopausal (no menses for ≥2 years), (2) surgically sterile (history of bilateral oophorectomy or hysterectomy), (3) women of childbearing potential with a documented negative serum or urine pregnancy test within 24 hours prior to 18F-FES administration, and who agree to use effective contraception during the trial.
* Subjects with serious and/or uncontrolled and/or unstable medical conditions (e.g., congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic kidney disease, or chronic liver disease)
* Subjects who are relatives or students of the investigator, or otherwise in a dependent relationship with the investigator
* Subjects who, in the judgment of the investigator, are unable to provide complete data for the clinical trial due to personal circumstances or other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient based detection rate of qualitative [18F]FES PET/CT evaluation for distant metastases | Baseline (index [18F]FES PET/CT image interpretation performed within 1 week after PET/CT acquisition, prior to initiation of definitive treatment)

SECONDARY OUTCOMES:
Patient-based sensitivity and specificity of qualitative [18F]FES PET/CT evaluation for distant metastases | From baseline [18F]FES PET/CT to confirmation of reference standard, assessed up to 6 months (histopathologic confirmation or clinical and imaging follow-up ≥6 months, through multidisciplinary consensus review)
Patient-based detection rate of qualitative [18F]FES PET/CT evaluation for cN3 lymph node metastases | Baseline (index [18F]FES PET/CT image interpretation performed within 1 week after PET/CT acquisition, prior to initiation of definitive treatment)
Patient-based sensitivity and specificity of qualitative [18F]FES PET/CT evaluation for cN3 lymph node metastases | From baseline [18F]FES PET/CT to confirmation of reference standard, assessed up to 6 months (histopathologic confirmation or clinical and imaging follow-up ≥6 months, through multidisciplinary consensus review)
Patient-based change rate in clinical management based on qualitative 18F-FES PET/CT evaluation | From baseline clinical management plan (pre-[18F]FES PET/CT) to final treatment decision after [18F]FES PET/CT, assessed within 4 weeks after PET/CT
Comparative patient-based evaluation of qualitative [18F]FES PET/CT and [18F]FDG PET/CT for detection rate of distant and cN3 lymph node metastases, and rate of change in clinical management | Baseline (paired [18F]FES PET/CT and [18F]FDG PET/CT image interpretation performed within 1 week after each PET/CT acquisition)
Comparative patient-based evaluation of qualitative [18F]FES PET/CT and [18F]FDG PET/CT for sensitivity, specificity of distant and cN3 lymph node metastases, and rate of change in clinical management | From baseline PET/CT imaging to confirmation of reference standard, assessed up to 6 months (histopathologic confirmation or clinical and imaging follow-up ≥6 months)

OTHER OUTCOMES:
Correlation between qualitative/quantitative [18F]FES PET/CT evaluation and response to neoadjuvant chemotherapy | From baseline [18F]FES PET/CT to post-surgical pathologic response assessment after completion of neoadjuvant chemotherapy, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyehyun Jeong, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No